CLINICAL TRIAL: NCT02403700
Title: Ridge Alterations Following Single Tooth Extraction in the Anterior Maxilla - A Prospective Clinical Study
Brief Title: Dimensional Soft and Hard Tissue Alterations Following Single Tooth Extraction in the Anterior Maxilla - A Prospective Clinical Study
Acronym: Alterations
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: ITI Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: 079/09; Grant No. 624_2009 (Other: ITI Foundation, Basel, Switzerland)
Record Dates: First submitted 2015-03-19; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Dimensional Alterations
Keywords: bone remodeling; bone resorption; three-dimensional imaging; clinical trial; dental implant; maxilla; bone healing
MeSH Terms: conditions — Bone Resorption | interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: One group observation study
  Interventions: Device: Cone beam computed tomography (CBCT)

INTERVENTIONS:
Device: Cone beam computed tomography (CBCT) — Dimensional changes are documented over a healing period of 8-weeks following single tooth extraction. To document these changes over time, two methods will be applied. Firstly, two cone beam computed tomographies (CBCT) will be obtained, one directly after tooth extraction, the other one at 8 weeks of socket healing prior to implant placement. The two CBCT's will be analyzed with a novel software program (InVivo Dental). Secondly, consecutive impressions will be made at day 0 (day of extraction), day 14, 28, 42, and 56 to digitally produce virtual 3D study models. These models can be analyzed with another software program (Geomagic Studi 10) to document the variations of the soft tissue in the extraction site.

SUMMARY:
Bone modeling after tooth extraction has a major consequence on implant therapy, in particular in the esthetic zone. In esthetic sites, no tissue loss should occur if an optimal esthetic outcome is expected. Recent experimental studies in dogs have shown that neither an immediate implant insertion nor ridge preservation techniques can prevent this bone modeling process.

DETAILED DESCRIPTION:
Background

The alveolar process is a tooth dependent tissue and develops in conjunction with the eruption of teeth. The size and the form of the tooth, the axis of eruption and eventual inclination determine the local volume as well as the shape of the alveolar process. It has been shown that after removing all teeth in humans, the alveolar ridge undergoes a process of resorption and atrophy.

In a recent animal study, Cardaropoli et al. (2003) assessed the healing events occurring in the extraction socket following tooth removal. The findings of this study demonstrated that the healing of an extraction socket involved a series of events including the formation of a coagulum that was replaced by a provisional connective tissue matrix, woven bone and lamellar bone and bone marrow. On day 30, mineralized bone occupied 88% of the socket volume. Hard tissue formation had started already after 2 weeks of healing, and then, after a month, the socket was filled with woven bone. Later, the woven bone was gradually replaced by lamellar bone and bone marrow. After 3 months of healing, a hard tissue bridge was consistently found to cover the crestal portion of the extraction site, which was formed by woven bone and lamellar bone. Araújo et al. (2005) analysed in an experimental study in dogs the ridge alterations following the extraction of premolars in the mandible. The authors observed that the resorption of the buccal and lingual walls occurred in two overlapping phases. Phase 1: The bundle bone - that lost its function and blood supply - was resorbed and replaced with woven bone. Vertical resorption was considerably greater on the buccal aspect of the alveolar crest, since this bone wall was much thinner then the lingual wall and was primarily comprised of bundle bone. Phase 2: An additional resorption occurred from the outer surfaces of both bone walls. The reason for this additional resorption has not been clearly ascertained. The hypothesis could be: Impaired superficial vascularisation by raising a mucoperiosteal flap; adjusting to the lack of continuous function; or the reestablishment of the ridge shape, which is genetically determined in the absence of teeth. A recent animal study confirmed that flap elevation plays an important role for a more pronounced superficial bone resorption following extraction , therefore, it seems critical that tooth extraction should be carried out without elevation of a mucoperiosteal flap. Even ridge preservation techniques are not able to prevent the contour changes after tooth extraction.

Objective

The aim of the present clinical study is to examine the dimensional changes of the alveolar ridge following single tooth extraction in the anterior maxilla of patients, in particular on the facial aspect of the alveolar ridge. These horizontal and vertical changes will be sequentially documented up to 8 weeks of healing before an implant is inserted using the concept of early implant placement. The study will also provide information about the anatomic situation of the facial bone wall in the anterior maxilla at the time of extraction, and the prevalence and extent of bone deficiencies on the facial aspect, when teeth need to be extracted.

Methods

To document these changes over time, two methods will be applied. Firstly, two cone beam computed tomographies (CBCT) will be obtained, one directly after tooth extraction, the other one at 8 weeks of socket healing prior to implant placement. The two CBCT's will be analyzed with a novel software program (InVivo Dental). Secondly, consecutive impressions will be made at day 0 (day of extraction), day 14, 28, 42, and 56 to digitally produce virtual 3D study models. These models can be analyzed with another software program (Geomagic) to document the variations of the soft tissue in the extraction site.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 18 years or older
* Absence of significant medical conditions
* Patients with healthy or effectually treated periodontal conditions
* Candidate for single tooth replacement in the anterior maxilla

Exclusion Criteria

* General contraindications for dental and/or surgical treatments
* Concurrent or previous immunosuppressant, bisphosphonate or high dose corticosteroid therapy
* Inflammatory and autoimmune disease of oral cavity
* Uncontrolled diabetes
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The group is selected from the referred patient pool. Age 18 or older. Absence of significant medical conditions. Sites with a need for single tooth extraction in the anterior maxilla.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in bone loss | 2-, 4-, 6-, 8-weeks
  Measured by segmented surface model superimpositions. Changes in bone loss between baseline and 8 week healing period using CBCT technology. From the Digital Imaging and Communications in Medicine (DICOM) files two surface mesh model were generated, which were superimposed and the changes were subsequently analyzed.
Change from baseline in soft tissue loss | 2-, 4-, 6-, 8-weeks
  Changes in soft tissue loss at baseline, 2-, 4-, 6- and 8 weeks were analyzed be dental impressions, which were superimposed as well and the changes were analyzed.

SECONDARY OUTCOMES:
Correlation between baseline facial bone thickness and dimensional soft tissue alterations during healing. | At baseline and 8-weeks
  To measure correlation, the Spearman Rank Correlation Coefficient was calculated. Nonparametric models for longitudinal data were applied to analyze the impact of bone wall phenotype and healing period upon dimensional alterations.

CONTACTS AND LOCATIONS:
Overall Officials: Chappuis, Principal Investigator — Dep. Oral surgery and Stomatology, University of Bern
Locations (1):
- Dep. of Oral Sugery and Stomatology, University of Bern, Canton of Bern, Switzerland

REFERENCES:
- [Result] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Result] Cardaropoli G, Araujo M, Lindhe J. Dynamics of bone tissue formation in tooth extraction sites. An experimental study in dogs. J Clin Periodontol. 2003 Sep;30(9):809-18. doi: 10.1034/j.1600-051x.2003.00366.x. PMID 12956657
- [Result] Araujo MG, Sukekava F, Wennstrom JL, Lindhe J. Tissue modeling following implant placement in fresh extraction sockets. Clin Oral Implants Res. 2006 Dec;17(6):615-24. doi: 10.1111/j.1600-0501.2006.01317.x. PMID 17092218
- [Result] Araujo MG, Lindhe J. Ridge alterations following tooth extraction with and without flap elevation: an experimental study in the dog. Clin Oral Implants Res. 2009 Jun;20(6):545-9. doi: 10.1111/j.1600-0501.2008.01703.x. PMID 19515033
- [Result] Januario AL, Duarte WR, Barriviera M, Mesti JC, Araujo MG, Lindhe J. Dimension of the facial bone wall in the anterior maxilla: a cone-beam computed tomography study. Clin Oral Implants Res. 2011 Oct;22(10):1168-1171. doi: 10.1111/j.1600-0501.2010.02086.x. Epub 2011 Feb 15. PMID 21320168
- [Result] Fickl S, Zuhr O, Wachtel H, Bolz W, Huerzeler M. Tissue alterations after tooth extraction with and without surgical trauma: a volumetric study in the beagle dog. J Clin Periodontol. 2008 Apr;35(4):356-63. doi: 10.1111/j.1600-051X.2008.01209.x. PMID 18353082
- [Result] Fickl S, Zuhr O, Wachtel H, Bolz W, Huerzeler MB. Hard tissue alterations after socket preservation: an experimental study in the beagle dog. Clin Oral Implants Res. 2008 Nov;19(11):1111-8. doi: 10.1111/j.1600-0501.2008.01575.x. PMID 18983313
- [Result] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Derived] Chappuis V, Engel O, Shahim K, Reyes M, Katsaros C, Buser D. Soft Tissue Alterations in Esthetic Postextraction Sites: A 3-Dimensional Analysis. J Dent Res. 2015 Sep;94(9 Suppl):187S-93S. doi: 10.1177/0022034515592869. Epub 2015 Jun 30. PMID 26130259